CLINICAL TRIAL: NCT02669017
Title: A Phase 1 Dose-escalation Study to Evaluate the Tolerability, Safety, Pharmacokinetics, and Antitumor Activity of ADCT-402 in Patients With Relapsed or Refractory B-cell Lineage Non Hodgkin Lymphoma (B-NHL)
Brief Title: Study of ADCT-402 in Patients With Relapsed or Refractory B-cell Lineage Non Hodgkin Lymphoma (B-NHL)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ADC Therapeutics S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADCT-402-101; 2016-000952-92 (EudraCT Number)
Record Dates: First submitted 2016-01-21; First posted 2016-01-29 (Estimated); Results first posted 2020-04-13 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Non-Hodgkin Lymphoma; Burkitt's Lymphoma; Chronic Lymphocytic Leukemia; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, Marginal Zone; Waldenstrom Macroglobulinemia; Primary Mediastinal B-cell Lymphoma
Keywords: Loncastuximab tesirine
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Burkitt Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma; Waldenstrom Macroglobulinemia | interventions — loncastuximab tesirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1: ADCT-402 dose escalation (Experimental): In Part 1 (dose escalation) participants will receive intravenous (IV) infusions of ADCT-402 at escalating doses, according to a 3+3 study design. Doses will be escalated from 15 µg/kg to 200 µg/kg on Day 1 of each cycle, with cycle lengths of 3 or 6 weeks.
  Interventions: Drug: ADCT-402
- Part 2: ADCT-402 dose expansion (Experimental): In Part 2 (expansion), participants will be assigned to the recommended dose level(s) and schedule(s) of ADCT-402 identified in Part 1 by the Dose Escalation Steering Committee.
  Participants will receive intravenous (IV) infusions of ADCT-402 at either 120 μg/kg or 150 μg/kg on Day 1 of each 3 week cycle (Q3W).
  Interventions: Drug: ADCT-402

INTERVENTIONS:
Drug: ADCT-402 — intravenous infusion
  Other Names: Loncastuximab tesirine; Zynlonta

SUMMARY:
This study evaluates ADCT-402 in participants with Relapsed or Refractory B-cell Lineage Non Hodgkin Lymphoma (B-NHL). Participants will participate in a dose escalation phase (Part 1) and dose expansion (Part 2). In Part 2, participants will receive the dose level identified in Part 1.

DETAILED DESCRIPTION:
Study ADCT-402-101 is the first clinical study with ADCT-402 in participants with B-cell Non Hodgkin Lymphoma (NHL).

ADCT-402 is an antibody drug conjugate (ADC) composed of a humanized antibody directed against human cluster of differentiation 19 (CD19), stochastically conjugated via a valine-alanine cleavable, maleimide linker to a pyrrolobenzodiazepine (PBD) dimer cytotoxin.

The study will be conducted in 2 parts. In Part 1 (dose escalation) participants will receive infusions of ADCT-402, at escalating doses. Part 1 will continue until the maximum tolerated dose is determined. In Part 2 (expansion), participants will be assigned to the recommended dose level(s) and schedule(s) of ADCT-402 identified in Part 1 by the Dose Escalation Steering Committee.

For each participant, the study will include a screening period (up to 28 days), a treatment period (until withdrawal), and a follow-up period to assess disease progression and survival for up to 12 months after the last dose of study drug. The total study duration will be dependent on overall participant tolerability to the study drug and response to treatment. It is anticipated that the duration of the entire study (Parts 1 and 2) could be approximately 3 years from first participant treated to last participant completed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants, ages 18 years or older with pathologically confirmed relapsed or refractory B-cell lineage NHL who have failed or are intolerant to established therapy, or for whom no other treatment options are available.
* Refractory or relapsed B-cell NHL (per World health Organization [WHO] Classification system).
* Availability of formalin-fixed paraffin-embedded (FFPE) tumor tissue block.
* Measurable disease, as defined by the 2014 Lugano Classification.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.
* Absolute neutrophil count (ANC) ≥1000/μL.
* Platelet count of ≥75000/μL.
* Hemoglobin ≥9.0 g/dL without transfusion within the 2 weeks prior to Day 1.
* Serum/plasma creatinine ≤1.5 mg/dL.
* Serum/plasma alkaline phosphatase, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) ≤2 times the upper limit of normal (ULN); ≤ 5 times ULN if there is liver or bone involvement.
* Total serum/plasma bilirubin ≤1.5 times ULN.
* Negative blood or urine beta-human chorionic gonadotropin (β-HCG) pregnancy test within 7 days prior to Day 1 for women of childbearing potential.
* Males, and female participants who are biologically capable of having children, must agree to use a medically acceptable method of birth control.

Exclusion Criteria:

* Participants who have any option for other treatment for B-cell NHL at the current state of disease.
* Active graft-versus-host disease.
* Autologous or allogenic transplant within the 60 days prior to the Screening visit.
* Known history of immunogenicity or hypersensitivity to a CD19 antibody.
* Evidence of myelodysplasia or myeloid leukemia by morphology, immunostains, flow cytometry, or cytogenetics on a bone marrow aspirate or biopsy.
* Known history of positive serum human ADA.
* Active autoimmune disease, motor neuropathy considered of autoimmune origin, and other central nervous system (CNS) autoimmune disease.
* Known seropositive for human immunodeficiency (HIV) virus, hepatitis B surface antigen (HbsAg), or antibody to hepatitis C virus (anti-HCV).
* History of Steven's Johnson's syndrome or toxic epidermal necrolysis syndrome.
* Pregnant or breastfeeding women.
* Significant medical comorbidities, including uncontrolled hypertension (diastolic blood pressure greater than 115 mm Hg), unstable angina, congestive heart failure (greater than New York Heart Association class II), severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia, poorly controlled diabetes, severe chronic pulmonary disease, coronary angioplasty, or myocardial infarction within 6 months prior to screening, or uncontrolled atrial or ventricular cardiac arrhythmias.
* Use of any other experimental medication(s) within 14 days or 5 half-lives but in no case less than 14 days prior to start of study treatment on Cycle 1, Day 1, except if approved by Sponsor.
* Steroid use equivalent to greater than 20 mg of prednisone within 4 weeks (28 days) prior to Day 1.
* Major surgery, chemotherapy, systemic therapy (excluding steroids hydroxyurea steroids, and any targeted small molecules or biologics), or radiotherapy, within 14 days or 5 half-lives (whichever is shorter) prior to Cycle 1, Day 1 treatment, except if approved by the Sponsor.
* Failure to recover (to Common Terminology Criteria for Adverse Events [CTCAE] Grade 0 or Grade 1) from acute non hematologic toxicity (except all grades alopecia or Grade 2 or lower neuropathy), due to previous therapy, prior to Screening.
* Congenital long QT syndrome or a corrected QTc interval ≥450 ms at the Screening visit.
* Active second primary malignancy other than non-melanoma skin cancers, non-metastatic prostate cancer, in situ cervical cancer, ductal or lobular carcinoma in situ of the breast, or other malignancy determined not be exclusionary.
* Any other significant medical illness, abnormality, or condition that would make the participant inappropriate for study participation or put the participant at risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2016-03; Primary Completion 2019-02-21 (Actual); Study Completion 2019-02-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (8):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Blood and Marrow Transplant Group of Georgia, Atlanta, Georgia
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Medical Center Herbert Irving Pavilion, New York, New York
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Greenville Health System, Institute for Translational Oncology Research, Clinical Research Unit, Greenville, South Carolina
  - Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin
- U.O Oncologia e Ematologia - Istituto Clinico Humanitas, Milan, Italy
- United Kingdom (2):
  - University College London Hospitals, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hess B, Townsend W, Ai W, Stathis A, Solh M, Alderuccio JP, Ungar D, Liao S, Liao L, Khouri L, Zhang X, Boni J. Efficacy and Safety Exposure-Response Analysis of Loncastuximab Tesirine in Patients with B cell non-Hodgkin Lymphoma. AAPS J. 2021 Dec 10;24(1):11. doi: 10.1208/s12248-021-00660-3. PMID 34893942
- [Derived] Hamadani M, Radford J, Carlo-Stella C, Caimi PF, Reid E, O'Connor OA, Feingold JM, Ardeshna KM, Townsend W, Solh M, Heffner LT, Ungar D, Wang L, Boni J, Havenith K, Qin Y, Kahl BS. Final results of a phase 1 study of loncastuximab tesirine in relapsed/refractory B-cell non-Hodgkin lymphoma. Blood. 2021 May 13;137(19):2634-2645. doi: 10.1182/blood.2020007512. PMID 33211842
- [Derived] Kahl BS, Hamadani M, Radford J, Carlo-Stella C, Caimi P, Reid E, Feingold JM, Ardeshna KM, Solh M, Heffner LT, Ungar D, He S, Boni J, Havenith K, O'Connor OA. A Phase I Study of ADCT-402 (Loncastuximab Tesirine), a Novel Pyrrolobenzodiazepine-Based Antibody-Drug Conjugate, in Relapsed/Refractory B-Cell Non-Hodgkin Lymphoma. Clin Cancer Res. 2019 Dec 1;25(23):6986-6994. doi: 10.1158/1078-0432.CCR-19-0711. Epub 2019 Nov 4. PMID 31685491

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were screened at 11 sites in 3 countries.
Groups:
- Part 1: 15 μg/kg Q3W: Participants received an intravenous (IV) infusion of ADCT-402 (15 μg/kg) on Day 1 of each 3 week cycle (Q3W).
- Part 1: 30 μg/kg Q3W: Participants received an intravenous (IV) infusion of ADCT-402 (30 μg/kg) on Day 1 of each 3 week cycle (Q3W).
- Part 1: 60 μg/kg Q3W: Participants received an intravenous (IV) infusion of ADCT-402 (60 μg/kg) on Day 1 of each 3 week cycle (Q3W).
- Part 1: 90 μg/kg Q3W: Participants received an intravenous (IV) infusion of ADCT-402 (90 μg/kg) on Day 1 of each 3 week cycle (Q3W).
- Part 1: 120 μg/kg Q3W; Part 2: 120 μg/kg Q3W: Participants received an intravenous (IV) infusion of ADCT-402 (120 μg/kg) on Day 1 of each 3 week cycle (Q3W).
- Part 1: 150 μg/kg Q3W; Part 2: 150 μg/kg Q3W: Participants received an intravenous (IV) infusion of ADCT-402 (150 μg/kg) on Day 1 of each 3 week cycle (Q3W).
- Part 1: 200 μg/kg Q3W and Q6W: Participants received an intravenous (IV) infusion of ADCT-402 (200 μg/kg) on Day 1 of each 3 week cycle (Q3W). Following protocol amendment 5, treatment cycle length was increased to 6 weeks (Q6W).
Period: Overall Study
Arm/Group | Part 1: 15 μg/kg Q3W | Part 1: 30 μg/kg Q3W | Part 1: 60 μg/kg Q3W | Part 1: 90 μg/kg Q3W | Part 1: 120 μg/kg Q3W | Part 2: 120 μg/kg Q3W | Part 1: 150 μg/kg Q3W | Part 2: 150 μg/kg Q3W | Part 1: 200 μg/kg Q3W and Q6W
Started | 4 | 4 | 4 | 5 | 16 | 26 | 19 | 69 | 36
Completed | 3 | 2 | 2 | 1 | 4 | 7 | 8 | 7 | 11
Not Completed | 1 | 2 | 2 | 4 | 12 | 19 | 11 | 62 | 25
Not completed — Death | 1 | 2 | 2 | 3 | 8 | 18 | 10 | 47 | 20
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Miscellaneous | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 13 | 2

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: 15 μg/kg Q3W | Part 1: 30 μg/kg Q3W | Part 1: 60 μg/kg Q3W | Part 1: 90 μg/kg Q3W | Part 1: 120 μg/kg Q3W | Part 2: 120 μg/kg Q3W | Part 1: 150 μg/kg Q3W | Part 2: 150 μg/kg Q3W | Part 1: 200 μg/kg Q3W and Q6W | Total
Number analyzed (Participants) | 4 | 4 | 4 | 5 | 16 | 26 | 19 | 69 | 36 | 183
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 3 | 2 | 3 | 14 | 13 | 43 | 19 | 99
  >=65 years | 3 | 3 | 1 | 3 | 13 | 12 | 6 | 26 | 17 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.5 (8.39) | 68.3 (11.53) | 51.3 (18.82) | 68.2 (12.38) | 71.0 (10.20) | 63.7 (13.37) | 58.5 (13.96) | 58.7 (15.82) | 61.7 (12.82) | 61.7 (14.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 3 | 3 | 7 | 6 | 34 | 10 | 69
  Male | 2 | 2 | 2 | 2 | 13 | 19 | 13 | 35 | 26 | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 1 | 6
  Not Hispanic or Latino | 4 | 4 | 4 | 5 | 16 | 25 | 18 | 65 | 35 | 176
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 4 | 4 | 4 | 4 | 14 | 19 | 19 | 61 | 35 | 164
  Race: Black or African American | 0 | 0 | 0 | 1 | 1 | 4 | 0 | 5 | 0 | 11
  Race: Asian | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 3
  Race: American Indian or Alaskan Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Race: Native Hawaiian or Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Race: Other | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 3
  Race: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Height [Mean (Standard Deviation); unit: cm] — Population: Height data was not collected for 2 participants because of complications during the collection of baseline measurements.
  cm
    number analyzed (Participants) | 4 | 4 | 4 | 5 | 16 | 26 | 19 | 68 | 35 | 181
    (all) | 172.23 (18.438) | 170.73 (12.545) | 173.65 (11.544) | 167.68 (10.275) | 170.72 (8.977) | 171.47 (9.790) | 172.79 (10.584) | 170.56 (11.908) | 171.29 (12.193) | 171.11 (11.221)
Weight [Mean (Standard Deviation); unit: kg] | 73.65 (7.204) | 78.73 (25.445) | 79.95 (26.942) | 86.38 (23.597) | 86.89 (25.996) | 78.66 (18.113) | 88.67 (20.820) | 77.87 (22.453) | 88.71 (24.834) | 82.23 (22.635)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: BMI could not be calculated for 2 participants due to missing height information.
  kg/m^2
    number analyzed (Participants) | 4 | 4 | 4 | 5 | 16 | 26 | 19 | 68 | 35 | 181
    (all) | 25.21 (3.971) | 26.60 (5.466) | 25.89 (5.428) | 30.77 (8.931) | 29.40 (6.882) | 26.68 (5.458) | 29.57 (5.575) | 26.62 (6.648) | 30.15 (7.235) | 27.93 (6.587)
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants]
  0: Fully Active | 2 | 0 | 2 | 0 | 7 | 7 | 4 | 20 | 12 | 54
  1: Restricted in Physical Activity; Ambulatory | 1 | 3 | 2 | 4 | 8 | 19 | 12 | 36 | 21 | 106
  2: Ambulatory and Capable of All Self-care | 1 | 1 | 0 | 1 | 1 | 0 | 2 | 12 | 3 | 21
  3: Capable of Only Limited Self-care | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
  4: Completely Disabled | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  5: Dead | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Dose-Limiting Toxicities (DLTs)
Description: A DLT is defined as any of the following events, except those that are clearly due to underlying disease or extraneous causes:
  A hematologic DLT is defined as:
  * CTCAE Grade 3 or 4 febrile neutropenia or neutropenic infection.
  * CTCAE Grade 4 neutropenia lasting >7 days.
  * CTCAE Grade 4 thrombocytopenia.
  * CTCAE Grade 3 thrombocytopenia with clinically significant bleeding, or Grade 3 thrombocytopenia requiring a platelet transfusion.
  * CTCAE Grade 4 anemia.
  A non-hematologic DLT is defined as:
  * CTCAE Grade 4 tumor lysis syndrome (TLS). Grade 3 TLS will not constitute DLT unless it leads to irreversible end-organ damage.
  * CTCAE Grade 3 or higher AE (including nausea, vomiting, diarrhea, and electrolyte imbalances lasting more than 48 hours despite optimal therapy; excluding all grades of alopecia).
  * CTCAE Grade 3 or higher hypersensitivity reaction (regardless of premedication).
  * CTCAE Grade 2 or higher skin ulceration.
Time Frame: Q3W schedule: Day 1 to End of Cycle 1 (3 weeks); Q6W schedule: Day 1 to End of Cycle 1 (6 weeks)
Population: All participants in Part 1 who completed at least one cycle of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: 15 μg/kg Q3W | Part 1: 30 μg/kg Q3W | Part 1: 60 μg/kg Q3W | Part 1: 90 μg/kg Q3W | Part 1: 120 μg/kg Q3W | Part 1: 150 μg/kg Q3W | Part 1: 200 μg/kg Q3W and Q6W
Number analyzed (Participants) | 4 | 4 | 3 | 5 | 16 | 16 | 25
Participants | 0 | 0 | 0 | 0 | 1 | 1 | 2

2. Primary Outcome: Recommended Dose of ADCT-402 for Part 2
Description: The recommended dose was established by the dose escalation steering committee and based on safety findings during Part 1 of the study.
Time Frame: Q3W schedule: Day 1 to End of Cycle 1 (3 weeks); Q6W schedule: Day 1 to End of Cycle 1 (6 weeks)
Population: All participants in Part 1 who completed at least one cycle of treatment.
Measure: Number; unit: μg/kg
Groups:
- Part 1: ADCT-402 Dose Escalation: In Part 1 (dose escalation) participants received intravenous (IV) infusions of ADCT-402, at escalating doses according to a 3+3 study design. Doses assessed:
  * Dose Level 1: 15 μg/kg on Day 1 of each 3 week cycle (Q3W)
  * Dose Level 2: 30 μg/kg Day 1 Q3W
  * Dose Level 3: 60 μg/kg Day 1 Q3W
  * Dose Level 4: 90 μg/kg Day 1 Q3W
  * Dose Level 5: 120 μg/kg Day 1 Q3W
  * Dose Level 6: 150 μg/kg Day 1 Q3W
  * Dose Level 7: 200 μg/kg Day 1 Q3W and on Day 1 of each 6 week cycle (Q6W).
Arm/Group | Part 1: ADCT-402 Dose Escalation
Number analyzed (Participants) | 73
μg/kg
  Recommended Part 2 Dose 1 | 120
  Recommended Part 2 Dose 2 | 150

3. Primary Outcome: Number of Participants Reporting at Least One Treatment Emergent Adverse Event (TEAE)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participants enrolled into this study regardless of its causal relationship to study drug. A TEAE is defined as any event not present before exposure to study drug or any event already present that worsens in either intensity or frequency after exposure to study drug.
Time Frame: Day 1 to End of Study (a maximum of 18 months)
Population: All participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: 15 μg/kg Q3W | Part 1: 30 μg/kg Q3W | Part 1: 60 μg/kg Q3W | Part 1: 90 μg/kg Q3W | Part 1: 120 μg/kg Q3W | Part 2: 120 μg/kg Q3W | Part 1: 150 μg/kg Q3W | Part 2: 150 μg/kg Q3W | Part 1: 200 μg/kg Q3W and Q6W
Number analyzed (Participants) | 4 | 4 | 4 | 5 | 16 | 26 | 19 | 69 | 36
Participants | 4 | 3 | 4 | 5 | 16 | 26 | 19 | 68 | 36

4. Primary Outcome: Number of Participants Reporting at Least One Treatment Emergent Serious Adverse Event (SAE)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant enrolled into this study regardless of its causal relationship to study drug. A treatment emergent AE (TEAE) is defined as any event not present before exposure to study drug or any event already present that worsens in either intensity or frequency after exposure to study drug. An SAE is defined as any event that results in death, is immediately life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect.
Time Frame: Day 1 to End of Study (a maximum of 18 months)
Population: All participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: 15 μg/kg Q3W | Part 1: 30 μg/kg Q3W | Part 1: 60 μg/kg Q3W | Part 1: 90 μg/kg Q3W | Part 1: 120 μg/kg Q3W | Part 2: 120 μg/kg Q3W | Part 1: 150 μg/kg Q3W | Part 2: 150 μg/kg Q3W | Part 1: 200 μg/kg Q3W and Q6W
Number analyzed (Participants) | 4 | 4 | 4 | 5 | 16 | 26 | 19 | 69 | 36
Participants | 1 | 1 | 0 | 4 | 4 | 14 | 6 | 40 | 15

5. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR was defined as the number of participants with a best overall response of complete response (CR) or partial response (PR) at the time each participant discontinued treatment with ADCT-402, before the start of subsequent anticancer therapy or procedure. Tumor response was assessed using the 2014 Lugano Classification for response.
  CR is defined as achieving either of the following:
  * Complete metabolic response.
  * Complete radiologic response (target node regress to <1.5 cm, no nonmeasured lesions, no organ enlargement, no new lesions and normal bone marrow morphology).
  PR is defined as achieving either of the following:
  * Partial metabolic response (findings indicate residual disease).
  * Partial remission (>50% decrease in target measurable nodes, regression/ absence/ no increase of nonmeasured lesions, spleen regressed by >50% in length and no new lesions).
Time Frame: Baseline to End of Study (a maximum of 18 months)
Population: All participants who received at least one dose of study treatment with a valid baseline disease assessment and at least one valid post-baseline disease assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: 15 μg/kg Q3W | Part 1: 30 μg/kg Q3W | Part 1: 60 μg/kg Q3W | Part 1: 90 μg/kg Q3W | Part 1: 120 μg/kg Q3W | Part 2: 120 μg/kg Q3W | Part 1: 150 μg/kg Q3W | Part 2: 150 μg/kg Q3W | Part 1: 200 μg/kg Q3W and Q6W
Number analyzed (Participants) | 4 | 4 | 4 | 5 | 16 | 26 | 19 | 68 | 34
Participants | 1 | 1 | 1 | 2 | 9 | 11 | 12 | 25 | 20

6. Secondary Outcome: Duration of Response (DoR)
Description: DoR is defined among responders (complete response [CR] and partial response [PR]) as the time from the earliest date of first response until the first date of either disease progression or death due to any cause. Tumor response was assessed using the 2014 Lugano Classification for response.
  Disease progression is defined as progressive metabolic disease or one of the follow:
  * Target node progression.
  * An individual extranodal lesion must be abnormal with length >1.5cm and/or increase of length >50%.
  * New or clear progression of nonmeasured lesions.
  * Regrowth of previously resolved lesions or new nodes >1.5 cm in length.
  * New or recurrent bone marrow involvement.
  DoR is presented overall for all participants who received ADCT-402, as specified in protocol section 7.4.
Time Frame: Baseline to End of Study (a maximum of 18 months)
Population: All participants who received at least one dose of study treatment with a valid baseline disease assessment and at least one valid post-baseline disease assessment. Results are pooled for all arms as specified in the protocol.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Parts 1 and 2: ADCT-402: In Part 1 (dose escalation) participants received intravenous (IV) infusions of ADCT-402, at escalating doses according to a 3+3 study design. Doses assessed:
  * Dose Level 1: 15 μg/kg on Day 1 of each 3 week cycle (Q3W)
  * Dose Level 2: 30 μg/kg Day 1 Q3W
  * Dose Level 3: 60 μg/kg Day 1 Q3W
  * Dose Level 4: 90 μg/kg Day 1 Q3W
  * Dose Level 5: 120 μg/kg Day 1 Q3W
  * Dose Level 6: 150 μg/kg Day 1 Q3W
  * Dose Level 7: 200 μg/kg Day 1 Q3W and on Day 1 of each 6 week cycle (Q6W).
  In Part 2 (expansion), participants received intravenous (IV) infusions of ADCT-402 at either 120 μg/kg or 150 μg/kg on Day 1 of each 3 week cycle (Q3W).
Arm/Group | Parts 1 and 2: ADCT-402
Number analyzed (Participants) | 180
months | 5.36 [4.04 to NA] — Upper limit of the confidence interval was not reached.

7. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the first dose of study drug treatment until the date of death due to any cause.
  OS is presented overall for all participants who received ADCT-402, as specified in protocol section 7.4.
Time Frame: Baseline to End of Study (a maximum of 18 months)
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Parts 1 and 2: ADCT-402
Number analyzed (Participants) | 180
months | 8.25 [6.74 to 10.68]

8. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined among the efficacy population as the time from first dose of study drug until either disease progression or death due to any cause. Tumor response was assessed using the 2014 Lugano Classification for response.
  Disease progression is defined as progressive metabolic disease or one of the follow:
  * Target node progression.
  * An individual extranodal lesion must be abnormal with length >1.5cm and/or increase of length >50%.
  * New or clear progression of nonmeasured lesions.
  * Regrowth of previously resolved lesions or new nodes >1.5 cm in length.
  * New or recurrent bone marrow involvement.
  PFS is presented overall for all participants who received ADCT-402, as specified in protocol section 7.4.
Time Frame: Baseline to End of Study (a maximum of 18 months)
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Parts 1 and 2: ADCT-402
Number analyzed (Participants) | 180
months | 3.09 [2.66 to 4.24]

9. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) for ADCT-402
Description: Cmax for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199).
  Results for Part 1 and Part 2 have been pooled for the same dosage and schedule, as specified in the protocol.
Time Frame: Q3W schedule: Day 1 (pre-dose and 1 to 6 hours post-dose), and days 2, 3, 5, 8, 15 and 21 of Cycles 1 and 2 (3 weeks cycle); Q6W schedule: Day 1 (pre-dose and 1 to 6 hours post-dose), and days 2, 3, 5, 8, 15 and 21 of Cycles 1 and 2 (6 week cycle)
Population: Only participants with evaluable pharmacokinetic (PK) results were included in the analysis. Where data is not presented, the PK profiles were non-measurable or short-lived in duration; therefore, no analysis could be performed.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Parts 1 and 2: 120 μg/kg Q3W: Participants received an intravenous (IV) infusion of ADCT-402 (120 μg/kg) on Day 1 of each 3 week cycle (Q3W). Parts 1 and 2 are pooled for PK analysis as specified in the protocol.
- Parts 1 and 2: 150 μg/kg Q3W: Participants received an intravenous (IV) infusion of ADCT-402 (150 μg/kg) on Day 1 of each 3 week cycle (Q3W). Parts 1 and 2 are pooled for PK analysis as specified in the protocol.
- Part 1: 200 μg/kg Q3W: Participants received an intravenous (IV) infusion of ADCT-402 (200 μg/kg) on Day 1 of each 3 week cycle (Q3W). Analysis was performed separately for Q3W and Q6W treatment cycles as specified in the protocol.
- Part 1: 200 μg/kg Q6W: Participants received an intravenous (IV) infusion of ADCT-402 (200 μg/kg) on Day 1 of each 6 week cycle (Q6W). Analysis was performed separately for Q3W and Q6W treatment cycles as specified in the protocol.
Arm/Group | Part 1: 15 μg/kg Q3W | Part 1: 30 μg/kg Q3W | Part 1: 60 μg/kg Q3W | Part 1: 90 μg/kg Q3W | Parts 1 and 2: 120 μg/kg Q3W | Parts 1 and 2: 150 μg/kg Q3W | Part 1: 200 μg/kg Q3W | Part 1: 200 μg/kg Q6W
Number analyzed (Participants) | 4 | 4 | 4 | 5 | 42 | 88 | 14 | 22
ng/mL
  PBD conjugated Ab: Cycle 1 | 260 (85.5) | 404 (161) | 721 (481) | 1088 (748) | 2374 (1040) | 3416 (3093) | 3619 (688) | 3798 (1332)
  PBD conjugated Ab: Cycle 2: number analyzed (Participants) | 4 | 4 | 3 | 5 | 40 | 72 | 11 | 12
  PBD conjugated Ab: Cycle 2 | 398 (284) | 1971 (2566) | 864 (686) | 1416 (799) | 2573 (655) | 3776 (2738) | 4293 (1021) | 3178 (1733)
  total Ab: Cycle 1: number analyzed (Participants) | 4 | 4 | 4 | 5 | 41 | 88 | 14 | 22
  total Ab: Cycle 1 | 298 (83.7) | 542 (192) | 856 (475) | 1560 (1102) | 2829 (1257) | 4383 (4460) | 4185 (1308) | 4543 (1805)
  total Ab: Cycle 2: number analyzed (Participants) | 4 | 4 | 3 | 5 | 39 | 72 | 11 | 12
  total Ab: Cycle 2 | 447 (283) | 2906 (4034) | 1275 (1025) | 2422 (983) | 3142 (888) | 4798 (3334) | 5059 (1027) | 3834 (1913)
  SG3199: Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 1 | 4 | 28 | 4 | 16
  SG3199: Cycle 1 |  |  |  | 0.102 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 0.0372 (0.0208) | 0.0570 (0.0454) | 0.0479 (0.0381) | 0.0468 (0.0333)
  SG3199: Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 2 | 4 | 15 | 3 | 4
  SG3199: Cycle 2 |  |  |  | 0.0704 (0.0152) | 0.0403 (0.0116) | 0.0485 (0.0449) | 0.0293 (0.00329) | 0.0516 (0.0325)

10. Secondary Outcome: Time to Reach the Maximum Serum Concentration (Tmax) for ADCT-402
Description: Tmax for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199).
  Results for Part 1 and Part 2 have been pooled for the same dosage and schedule, as specified in the protocol.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Median (Full Range); unit: days
Arm/Group | Part 1: 15 μg/kg Q3W | Part 1: 30 μg/kg Q3W | Part 1: 60 μg/kg Q3W | Part 1: 90 μg/kg Q3W | Parts 1 and 2: 120 μg/kg Q3W | Parts 1 and 2: 150 μg/kg Q3W | Part 1: 200 μg/kg Q3W | Part 1: 200 μg/kg Q6W
Number analyzed (Participants) | 4 | 4 | 4 | 5 | 42 | 88 | 14 | 22
days
  PBD conjugated Ab: Cycle 1 | 0.0837 [0.0833 to 0.0854] | 0.0833 [0.0431 to 0.319] | 0.0819 [0.0417 to 0.0847] | 0.0500 [0.0417 to 0.0875] | 0.0833 [0.0403 to 0.296] | 0.0840 [0.0417 to 0.305] | 0.0858 [0.0417 to 0.285] | 0.0840 [0.0417 to 0.276]
  PBD conjugated Ab: Cycle 2: number analyzed (Participants) | 4 | 4 | 3 | 5 | 40 | 72 | 11 | 12
  PBD conjugated Ab: Cycle 2 | 0.122 [0.0660 to 0.170] | 0.0618 [0.0417 to 0.0875] | 0.0417 [0.0222 to 0.165] | 0.0833 [0.0229 to 0.0882] | 0.0830 [0.0208 to 0.278] | 0.0642 [0.0208 to 1.00] | 0.0854 [0.0208 to 1.00] | 0.0826 [0.0257 to 0.172]
  total Ab: Cycle 1: number analyzed (Participants) | 4 | 4 | 4 | 5 | 41 | 88 | 14 | 22
  total Ab: Cycle 1 | 0.0844 [0.0438 to 0.292] | 0.0833 [0.0431 to 0.0896] | 0.0833 [0.0806 to 0.0847] | 0.0500 [0.0417 to 0.169] | 0.0833 [0.0403 to 0.294] | 0.0837 [0.0403 to 0.299] | 0.0840 [0.0417 to 0.285] | 0.0837 [0.0417 to 0.271]
  total Ab: Cycle 2: number analyzed (Participants) | 4 | 4 | 3 | 5 | 39 | 72 | 11 | 12
  total Ab: Cycle 2 | 0.0649 [0.0431 to 0.0868] | 0.0618 [0.0417 to 0.0875] | 0.0417 [0.0222 to 0.0854] | 0.0833 [0.0229 to 0.159] | 0.0632 [0.0208 to 0.275] | 0.0639 [0 to 2.11] | 0.132 [0.0208 to 4.00] | 0.0858 [0.0257 to 0.172]
  SG3199: Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 1 | 4 | 28 | 4 | 16
  SG3199: Cycle 1 |  |  |  | 0.0833 [0.0833 to 0.0833] | 0.0854 [0.0458 to 0.172] | 0.0844 [0.0417 to 0.294] | 0.128 [0.0833 to 0.285] | 0.165 [0.0417 to 6.81]
  SG3199: Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 2 | 4 | 15 | 3 | 4
  SG3199: Cycle 2 |  |  |  | 1.05 [0.0417 to 2.06] | 0.120 [0.0840 to 0.153] | 0.0632 [0.0222 to 13.8] | 0.165 [0.0299 to 0.992] | 0.162 [0.0833 to 0.280]

11. Secondary Outcome: Area Under the Serum Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) for ADCT-402
Description: AUClast for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199).
  Results for Part 1 and Part 2 have been pooled for the same dosage and schedule, as specified in the protocol.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | Part 1: 15 μg/kg Q3W | Part 1: 30 μg/kg Q3W | Part 1: 60 μg/kg Q3W | Part 1: 90 μg/kg Q3W | Parts 1 and 2: 120 μg/kg Q3W | Parts 1 and 2: 150 μg/kg Q3W | Part 1: 200 μg/kg Q3W | Part 1: 200 μg/kg Q6W
Number analyzed (Participants) | 4 | 4 | 4 | 5 | 42 | 88 | 14 | 22
day*ng/mL
  PBD conjugated Ab: Cycle 1 | 1063 (1340) | 2390 (826) | 3875 (3228) | 6587 (6842) | 13544 (7503) | 14258 (8248) | 30571 (12425) | 30386 (16960)
  PBD conjugated Ab: Cycle 2: number analyzed (Participants) | 4 | 4 | 3 | 5 | 40 | 72 | 11 | 12
  PBD conjugated Ab: Cycle 2 | 1933 (2289) | 2955 (1132) | 5573 (4827) | 10369 (11656) | 18707 (10505) | 23109 (15370) | 48183 (20288) | 39609 (24852)
  total Ab: Cycle 1: number analyzed (Participants) | 4 | 4 | 4 | 5 | 41 | 88 | 14 | 22
  total Ab: Cycle 1 | 1185 (1540) | 3194 (1136) | 5032 (4334) | 8869 (9108) | 15980 (7649) | 16973 (9745) | 33834 (14888) | 36099 (20829)
  total Ab: Cycle 2: number analyzed (Participants) | 4 | 4 | 3 | 5 | 39 | 72 | 11 | 12
  total Ab: Cycle 2 | 1924 (2576) | 3986 (1725) | 7958 (6882) | 14025 (15704) | 23428 (13513) | 28657 (19457) | 57450 (26899) | 49892 (31012)
  SG3199: Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 1 | 4 | 28 | 4 | 16
  SG3199: Cycle 1 |  |  |  | 0.00213 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 0.00462 (0.00671) | 0.0222 (0.0423) | 0.0174 (0.0303) | 0.0436 (0.0959)
  SG3199: Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 2 | 4 | 15 | 3 | 4
  SG3199: Cycle 2 |  |  |  | 0.0242 (0.0234) | 0.154 (0.286) | 0.0108 (0.0248) | 0.00425 (0.00461) | 0.00332 (0.00215)

12. Secondary Outcome: Area Under the Serum Concentration-Time Curve From Time 0 to the End of the Dosing Interval (AUCtau) for ADCT-402
Description: AUCtau for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199).
  Results for Part 1 and Part 2 have been pooled for the same dosage and schedule, as specified in the protocol.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | Part 1: 15 μg/kg Q3W | Part 1: 30 μg/kg Q3W | Part 1: 60 μg/kg Q3W | Part 1: 90 μg/kg Q3W | Parts 1 and 2: 120 μg/kg Q3W | Parts 1 and 2: 150 μg/kg Q3W | Part 1: 200 μg/kg Q3W | Part 1: 200 μg/kg Q6W
Number analyzed (Participants) | 4 | 4 | 3 | 5 | 40 | 72 | 11 | 12
day*ng/mL
  PBD conjugated Ab: Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PBD conjugated Ab: Cycle 2: number analyzed (Participants) | 4 | 4 | 2 | 5 | 40 | 72 | 11 | 12
  PBD conjugated Ab: Cycle 2 | 2285 (2928) | 3458 (1426) | 10575 (1121) | 10171 (11244) | 19890 (8968) | 22859 (12080) | 39362 (9800) | 38466 (23514)
  total Ab: Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  total Ab: Cycle 2: number analyzed (Participants) | 4 | 4 | 3 | 4 | 39 | 72 | 11 | 12
  total Ab: Cycle 2 | 2636 (3387) | 4662 (2096) | 10211 (8827) | 17141 (15029) | 24247 (10902) | 28041 (15312) | 46469 (12675) | 48524 (28858)
  SG3199: Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SG3199: Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time 0 to Infinity (AUCinf) for ADCT-402
Description: AUCinf for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199).
  Results for Part 1 and Part 2 have been pooled for the same dosage and schedule, as specified in the protocol.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | Part 1: 15 μg/kg Q3W | Part 1: 30 μg/kg Q3W | Part 1: 60 μg/kg Q3W | Part 1: 90 μg/kg Q3W | Parts 1 and 2: 120 μg/kg Q3W | Parts 1 and 2: 150 μg/kg Q3W | Part 1: 200 μg/kg Q3W | Part 1: 200 μg/kg Q6W
Number analyzed (Participants) | 3 | 2 | 2 | 2 | 15 | 47 | 4 | 13
day*ng/mL
  PBD conjugated Ab: Cycle 1 | 432 (173) | 2001 (663) | 5333 (4002) | 5622 (7170) | 10232 (6220) | 11498 (8175) | 29174 (25838) | 32629 (19488)
  PBD conjugated Ab: Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  total Ab: Cycle 1: number analyzed (Participants) | 1 | 0 | 0 | 1 | 12 | 37 | 2 | 12
  total Ab: Cycle 1 | 869 (NA) — Standard deviation could not be determined as only one participant had evaluable data. |  |  | 16409 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 13292 (8495) | 12692 (8968) | 38991 (53597) | 43952 (24032)
  total Ab: Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SG3199: Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  SG3199: Cycle 1 |  |  |  |  |  | 0.154 (NA) — Standard deviation could not be determined as only one participant had evaluable data. |  |
  SG3199: Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Terminal Half-life (Thalf) of ADCT-402
Description: Thalf of Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199).
  Results for Part 1 and Part 2 have been pooled for the same dosage and schedule, as specified in the protocol.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Median (Full Range); unit: days
Arm/Group | Part 1: 15 μg/kg Q3W | Part 1: 30 μg/kg Q3W | Part 1: 60 μg/kg Q3W | Part 1: 90 μg/kg Q3W | Parts 1 and 2: 120 μg/kg Q3W | Parts 1 and 2: 150 μg/kg Q3W | Part 1: 200 μg/kg Q3W | Part 1: 200 μg/kg Q6W
Number analyzed (Participants) | 4 | 4 | 2 | 4 | 38 | 69 | 11 | 13
days
  PBD conjugated Ab: Cycle 1: number analyzed (Participants) | 3 | 2 | 2 | 2 | 15 | 47 | 4 | 13
  PBD conjugated Ab: Cycle 1 | 1.15 [1.04 to 2.56] | 6.84 [5.74 to 7.94] | 6.30 [4.30 to 8.30] | 3.97 [0.923 to 7.01] | 6.33 [0.515 to 9.50] | 6.43 [0.146 to 13.1] | 7.96 [6.43 to 16.6] | 10.4 [0.0560 to 19.6]
  PBD conjugated Ab: Cycle 2: number analyzed (Participants) | 4 | 4 | 2 | 4 | 38 | 69 | 11 | 12
  PBD conjugated Ab: Cycle 2 | 3.98 [0.909 to 11.1] | 10.1 [6.72 to 17.1] | 16.3 [11.1 to 21.4] | 11.4 [1.78 to 19.2] | 12.5 [1.74 to 28.7] | 11.6 [1.50 to 33.0] | 16.3 [8.14 to 28.8] | 15.5 [4.82 to 25.0]
  total Ab: Cycle 1: number analyzed (Participants) | 1 | 0 | 0 | 1 | 12 | 37 | 2 | 12
  total Ab: Cycle 1 | 2.75 [2.75 to 2.75] |  |  | 8.82 [8.82 to 8.82] | 7.00 [0.325 to 10.6] | 6.58 [0.0759 to 17.7] | 9.39 [0.661 to 18.1] | 12.7 [0.248 to 19.0]
  total Ab: Cycle 2: number analyzed (Participants) | 4 | 3 | 2 | 4 | 34 | 66 | 10 | 12
  total Ab: Cycle 2 | 3.71 [0.860 to 13.0] | 9.58 [7.11 to 15.4] | 16.5 [12.9 to 20.0] | 13.4 [1.27 to 38.5] | 14.9 [2.07 to 33.5] | 14.3 [0.269 to 36.0] | 14.7 [8.47 to 27.8] | 18.4 [6.18 to 39.9]
  SG3199: Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SG3199: Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Apparent Clearance (CL) at Steady State for ADCT-402
Description: CL of Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199).
  Results for Part 1 and Part 2 have been pooled for the same dosage and schedule, as specified in the protocol.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: liters/day
Arm/Group | Part 1: 15 μg/kg Q3W | Part 1: 30 μg/kg Q3W | Part 1: 60 μg/kg Q3W | Part 1: 90 μg/kg Q3W | Parts 1 and 2: 120 μg/kg Q3W | Parts 1 and 2: 150 μg/kg Q3W | Part 1: 200 μg/kg Q3W | Part 1: 200 μg/kg Q6W
Number analyzed (Participants) | 4 | 4 | 3 | 5 | 40 | 72 | 11 | 13
liters/day
  PBD conjugated Ab: Cycle 1: number analyzed (Participants) | 3 | 2 | 2 | 2 | 15 | 47 | 4 | 13
  PBD conjugated Ab: Cycle 1 | 2.49 (0.978) | 1.08 (0.164) | 0.696 (0.444) | 7.13 (8.91) | 2.09 (4.07) | 3.84 (8.53) | 3.11 (5.30) | 12.6 (39.4)
  PBD conjugated Ab: Cycle 2: number analyzed (Participants) | 4 | 4 | 2 | 5 | 40 | 72 | 11 | 12
  PBD conjugated Ab: Cycle 2 | 1.78 (1.80) | 0.646 (0.348) | 0.415 (0.205) | 19.6 (40.6) | 17.8 (109) | 0.986 (2.48) | 0.407 (0.143) | 0.349 (0.210)
  total Ab: Cycle 1: number analyzed (Participants) | 1 | 0 | 0 | 1 | 12 | 37 | 2 | 12
  total Ab: Cycle 1 | 1.28 (NA) — Standard deviation could not be determined as only one participant had evaluable data. |  |  | 0.640 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 2.47 (5.00) | 3.87 (8.95) | 7.12 (9.62) | 2.02 (5.11)
  total Ab: Cycle 2: number analyzed (Participants) | 4 | 4 | 3 | 4 | 39 | 72 | 11 | 12
  total Ab: Cycle 2 | 1.76 (1.71) | 0.577 (0.309) | 38.1 (65.5) | 1.42 (2.06) | 0.581 (0.660) | 1.05 (2.91) | 0.417 (0.161) | 0.323 (0.187)
  SG3199: Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  SG3199: Cycle 1 |  |  |  |  |  | 627 (NA) — Standard deviation could not be determined as only one participant had evaluable data. |  |
  SG3199: Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Volume of Distribution at Steady State (Vss) for ADCT-402
Description: Vss for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199).
  Results for Part 1 and Part 2 have been pooled for the same dosage and schedule, as specified in the protocol.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Part 1: 15 μg/kg Q3W | Part 1: 30 μg/kg Q3W | Part 1: 60 μg/kg Q3W | Part 1: 90 μg/kg Q3W | Parts 1 and 2: 120 μg/kg Q3W | Parts 1 and 2: 150 μg/kg Q3W | Part 1: 200 μg/kg Q3W | Part 1: 200 μg/kg Q6W
Number analyzed (Participants) | 4 | 4 | 2 | 4 | 38 | 69 | 11 | 13
liters
  PBD conjugated Ab: Cycle 1: number analyzed (Participants) | 3 | 2 | 2 | 2 | 15 | 47 | 4 | 13
  PBD conjugated Ab: Cycle 1 | 4.47 (0.759) | 10.3 (4.83) | 4.96 (0.318) | 9.68 (2.68) | 5.95 (1.86) | 7.59 (6.18) | 11.5 (11.1) | 7.18 (2.52)
  PBD conjugated Ab: Cycle 2: number analyzed (Participants) | 4 | 4 | 2 | 4 | 38 | 69 | 11 | 12
  PBD conjugated Ab: Cycle 2 | 3.82 (1.25) | 10.1 (8.57) | 8.29 (0.540) | 7.62 (1.09) | 6.71 (3.13) | 7.48 (4.29) | 9.18 (3.43) | 6.21 (1.70)
  total Ab: Cycle 1: number analyzed (Participants) | 1 | 0 | 0 | 1 | 12 | 37 | 2 | 12
  total Ab: Cycle 1 | 4.71 (NA) — Standard deviation could not be determined as only one participant had evaluable data. |  |  | 7.84 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 5.51 (1.29) | 6.60 (3.16) | 7.91 (0.0252) | 7.20 (2.03)
  total Ab: Cycle 2: number analyzed (Participants) | 4 | 3 | 2 | 4 | 34 | 66 | 10 | 12
  total Ab: Cycle 2 | 3.83 (0.854) | 9.62 (8.54) | 7.30 (1.38) | 8.52 (1.34) | 8.11 (4.57) | 8.21 (3.64) | 9.46 (5.26) | 6.86 (2.27)
  SG3199: Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  SG3199: Cycle 1 |  |  |  |  |  | 335 (NA) — Standard deviation could not be determined as only one participant had evaluable data. |  |
  SG3199: Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Accumulation Index (AI) for ADCT-402
Description: AI for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199). AI is the ratio of area under the serum concentration-time curve (AUC) from 0 to 21 days for Cycle 2 divided by AUC from 0 to 21 days for Cycle 1 (Q3W schedule: 3 week cycle length; Q6W schedule: 6 week cycle length). It is the increase in drug plasma concentration after multiple dosing until a steady state is reached.
  Results for Part 1 and Part 2 have been pooled for the same dosage and schedule, as specified in the protocol.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Part 1: 15 μg/kg Q3W | Part 1: 30 μg/kg Q3W | Part 1: 60 μg/kg Q3W | Part 1: 90 μg/kg Q3W | Parts 1 and 2: 120 μg/kg Q3W | Parts 1 and 2: 150 μg/kg Q3W | Part 1: 200 μg/kg Q3W | Part 1: 200 μg/kg Q6W
Number analyzed (Participants) | 4 | 4 | 2 | 4 | 38 | 69 | 11 | 12
ratio
  PBD conjugated Ab: Cycle 2 | 1.12 (0.173) | 1.37 (0.264) | 1.70 (0.467) | 1.42 (0.399) | 1.47 (0.369) | 1.46 (0.368) | 1.76 (0.385) | 1.23 (0.160)
  total Ab: Cycle 2: number analyzed (Participants) | 4 | 3 | 2 | 4 | 34 | 66 | 10 | 12
  total Ab: Cycle 2 | 1.15 (0.229) | 1.35 (0.252) | 1.71 (0.325) | 1.80 (0.962) | 1.62 (0.492) | 1.63 (0.486) | 1.78 (0.418) | 1.36 (0.314)
  SG3199: Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: Number of Participants With Anti-drug Antibody Response (ADA) Against ADCT-402
Description: Blood serum samples were collected and analysed to determine the presence or absence of ADA.
  ADA is presented overall for all participants who received ADCT-402, as specified in protocol section 7.4.
Time Frame: Q3W schedule: Day 1 to End of Cycle 1 (3 weeks); Q6W schedule: Day 1 to End of Cycle 1 (6 weeks)
Population: All participants who were tested for ADA.
Measure: Count of Participants; unit: Participants
Arm/Group | Parts 1 and 2: ADCT-402
Number analyzed (Participants) | 183
Participants
  Confirmed positive ADA pre-dose | 5
  Confirmed positive ADA post-dose only | 1
  Confirmed positive ADA at anytime | 6

ADVERSE EVENTS:
Time Frame: Day 1 to End of Study (a maximum of 18 months)
Arm/Group | Part 1: 15 μg/kg Q3W | Part 1: 30 μg/kg Q3W | Part 1: 60 μg/kg Q3W | Part 1: 90 μg/kg Q3W | Part 1: 120 μg/kg Q3W | Part 2: 120 μg/kg Q3W | Part 1: 150 μg/kg Q3W | Part 2: 150 μg/kg Q3W | Part 1: 200 μg/kg Q3W and Q6W
All-Cause Mortality (participants affected / at risk) | 1/4 | 2/4 | 2/4 | 3/5 | 8/16 | 18/26 | 10/19 | 47/69 | 20/36
Serious Adverse Events (participants affected / at risk) | 1/4 | 1/4 | 0/4 | 4/5 | 4/16 | 4/26 | 6/19 | 40/69 | 15/36
Other Adverse Events (participants affected / at risk) | 4/4 | 3/4 | 4/4 | 5/5 | 16/16 | 25/26 | 19/19 | 65/69 | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: 15 μg/kg Q3W (N=4) | Part 1: 30 μg/kg Q3W (N=4) | Part 1: 60 μg/kg Q3W (N=4) | Part 1: 90 μg/kg Q3W (N=5) | Part 1: 120 μg/kg Q3W (N=16) | Part 2: 120 μg/kg Q3W (N=26) | Part 1: 150 μg/kg Q3W (N=19) | Part 2: 150 μg/kg Q3W (N=69) | Part 1: 200 μg/kg Q3W and Q6W (N=36)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 5 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Abdominal compartment syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 8 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 2 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia haemophilus (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Progressive multifocal leukoencephalopathy (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oedema genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Perineal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Scrotal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: 15 μg/kg Q3W (N=4) | Part 1: 30 μg/kg Q3W (N=4) | Part 1: 60 μg/kg Q3W (N=4) | Part 1: 90 μg/kg Q3W (N=5) | Part 1: 120 μg/kg Q3W (N=16) | Part 2: 120 μg/kg Q3W (N=26) | Part 1: 150 μg/kg Q3W (N=19) | Part 2: 150 μg/kg Q3W (N=69) | Part 1: 200 μg/kg Q3W and Q6W (N=36)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 3 | 1 | 9 | 7 | 25 | 14
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 2 | 3 | 4 | 3 | 17 | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 3 | 6 | 3 | 13 | 9
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 3 | 3
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 2 | 1
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 5 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2
Visual impairment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 4 | 8 | 5 | 22 | 16
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2 | 9 | 2 | 18 | 6
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2 | 5 | 2 | 15 | 7
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 3 | 2 | 3 | 13 | 5
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2 | 6 | 4 | 7 | 7
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 4 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 5 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 2
Anal incontinence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 2 | 3 | 11 | 11 | 8 | 24 | 16
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 8 | 4 | 9 | 22 | 14
Pyrexia (General disorders) | 1 | 0 | 0 | 1 | 0 | 6 | 2 | 8 | 11
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 4
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 3 | 4
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 2 | 4
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 3
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 4 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 5 | 1
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 3
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Food allergy (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 7 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 3 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Corona virus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 2 | 3 | 4 | 7 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 2 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 4 | 4 | 9 | 3 | 19 | 17
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 3 | 1 | 5 | 2 | 16 | 9
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 2 | 1 | 4 | 1 | 14 | 11
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 7 | 3 | 11 | 11
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 2 | 1 | 5 | 3 | 11 | 9
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 1 | 3 | 3 | 5 | 8 | 8
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 5 | 2 | 4 | 9
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 6 | 6
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 2 | 3
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 2 | 3
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 3
Amylase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 1
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 2
Lipase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Blood bicarbonate increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1 | 6 | 2 | 11 | 12
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 3 | 12 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 3 | 3 | 7 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 5 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 8 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 6
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 3 | 3
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 4 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 3 | 1 | 1 | 3 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 4 | 3 | 5 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 7 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 4 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 4 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Limb mass (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 5 | 4 | 5 | 4
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 2 | 3 | 2 | 4 | 5
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 2
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 4 | 4
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 3
Breast oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 4 | 7 | 4 | 15 | 7
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 4 | 4 | 3 | 15 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3 | 7 | 2 | 14 | 8
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 2 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 3 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 3 | 4 | 8 | 19 | 9
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2 | 3 | 2 | 9 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 2 | 2 | 2 | 5 | 7
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 3 | 1 | 2 | 5 | 5
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 3 | 0 | 2 | 3 | 4
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 2 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 1 | 2 | 0 | 1 | 2
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 4
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 3
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 2 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 2 | 3 | 0 | 4 | 4
Hypotension (Vascular disorders) | 2 | 0 | 0 | 0 | 1 | 3 | 1 | 3 | 4
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 3 | 0
Bladder spasm (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI can publish after first multi-site publication, or if no multi-site publication is made within 18 months of study completion/termination. The only disclosure restriction on the PI is the sponsor can review results comms. prior to public release and can embargo comms. regarding trial results for a period that is more than 60 but less than or equal to 180 days from the time submitted to sponsor for review. The sponsor can't require changes to the communication and can't extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2017-10-16): https://cdn.clinicaltrials.gov/large-docs/17/NCT02669017/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-10): https://cdn.clinicaltrials.gov/large-docs/17/NCT02669017/SAP_001.pdf